CLINICAL TRIAL: NCT01238406
Title: Multicenter, Prospective, Open Label, Cross Over, Pilot Trial to Evaluate Blood Glucose Control Overnight Under Closed-loop Insulin Delivery With MD Logic Artificial Pancreas (MDLAP)System in Patients With Type 1 Diabetes
Brief Title: Overnight MD-Logic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: rmc006000ctil
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Closed loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD-logic Artificial Pancreas (MDLAP) system (Experimental): Use of the closed loop MD-logic Artificial Pancreas(MDLAP)System
  Interventions: Device: MD-logic Artificial Pancreas (MDLAP)
- Standard treatment with insulin pump (Active Comparator): Standard treatment with sensor augmented pump therapy
  Interventions: Device: Standard treatment with insulin pump

INTERVENTIONS:
Device: MD-logic Artificial Pancreas (MDLAP) — Treatment with the closed loop MD-logic Artificial Pancreas(MDLAP)System
  Arms: MD-logic Artificial Pancreas (MDLAP) system
Device: Standard treatment with insulin pump — Standard treatment with sensor augmented pump therapy
  Arms: Standard treatment with insulin pump

SUMMARY:
Study design: Multicenter,randomized, prospective, open label, cross over, six segments, pilot trial to evaluate blood glucose control overnight under closed-loop insulin delivery with MD-Logic Artificial Pancreas (MDLAP) system in patients with type 1 diabetes.

on the first segment 15 eligible subjects will be enrolled from the three participating centers (5 patients at each center). All 15 patients will participate in the overnight closed loop session in the hospital settings.

On the second segment, 54 eligible subjects will be enrolled (18 at each center). Each subject will participate in the two consecutive overnight sessions in diabetes camp settings, one under closed-loop with MDLAP and one under sensor augmented pump therapy.

In the third segment,9-20 eligible patients will be enrolled at the Israeli center only.Each subject will participate in up to four consecutive overnight under closed loop with MDLAP and up to four additional overnight under regular sensor augmented pump therapy at home.

On the fourth segment, 45-60 patients will be enrolled at the Israeli center only. This segment will be conducted at a diabetes camp and will consist of two main parts. In part 1, 15-20 patients will be randomized to participate in one of the two groups: 2-4 nights under closed loop control while the MD-Logic learning algorithm is activated or 2-4 nights under closed loop control without activating the MD-Logic learning algorithm. In part 2 of the forth segment 30-40 patients will participate in two consecutive24-48 hours sessions,one under closed loop control and the second under sensor augmented pump therapy.

On the fifth segment 40-80 eligible patients will be enrolled at the Israeli center only.The first 10 patients will participate in a pilot session and data gathered at this pilot session will not be used at the final analysis.This segment will consist of two parts. At part 1 each subject will participate in 4weeks-1.5 months period of over nights either using closed-loop with MDLAP or using sensor augmented pump (SAP) therapy.At the end of the first 4 weeks-1.5 months of the study, statistical analysis will be performed in order to decide whether to extend the study with an optional period of extra 4 weeks-1.5 months.In case it will be decided to extend the study, additional 4 weeks-1.5 months intervention period following completion of final visit activities will be offered to participants. Subjects that have participated in the control group (sensor augmented pump therapy) will be offered the opportunity to continue to 4 weeks-1.5 months of closed-loop control and the study group will be offered to switch to sensor augmented pump therapy. In segment 5 part 2, up to 40 patients will be enrolled. Each patient will participate in 3 months study period either using overnight closed loop under MDLAP or sensor augmented pump therapy.Participants in segment 5 part 2 will be offered to participate in part 2A. At this part, sleep quality assessment will be made (by using actigraf and sleep questionnaire) At the end of this period an optional 3 months extension period will be offered with the other arm (cross-over)

Segment 6 will be consist of two main parts.In part 1, up to 40 eligible patients will be enrolled at the Israeli center only. Each subject will participate in up to 72 hours of closed-loop with MDLAP at home and up to 72 hours under regular sensor augmented pump therapy . The sequence of the treatment intervention will be randomly assigned. The sequence of the treatment intervention will be randomly assigned. In part 2 of this segment 40 eligible patients will enrolled at the Israeli center only. Each subject will participate in up to 2 weeks of closed loop with MDLAP at home and up to 2 weeks under regular sensor augmented pump therapy. The sequence of the treatment intervention will be randomly assigned

Objectives: The objective of this feasibility study is to evaluate the safety and efficacy of blood glucose control using the MD-Logic Artificial Pancreas System in individuals with type 1 diabetes in the hospital settings,at a diabetes camp and finally at patient's home.

DETAILED DESCRIPTION:
In the last two decades, remarkable technological progress has been made with the development of continuous glucose sensors, miniature devices, implantable pumps and sensors and wireless communications, interest in the closed-loop insulin delivery was revived.

Control trails that evaluate the clinical benefits of continuous glucose sensor have shown improved HbA1c with no significant increase in sever hypoglycemia, trend towards lower hypoglycemic episodes although not significant and no significant change in sever hypoglycemia. One of the main drawbacks of continuous glucose sensor is noncompliant of the patient, the flow of information and the need to act accordingly makes this devise a burden for some patients. Theoretically subcutaneous insulin pumps and glucose sensors attached to an artificial pancreas in a closed-loop system can mimic the activity of functioning pancreatic beta cells, with strict control of blood glucose levels. Such a system may also offer an opportunity to free the patients from the daily burden of dealing with their diabetes.

We developed the MD-Logic Artificial Pancreas (MDLAP) which is based on a model which imitates the logic of diabetes care givers.

We aimed to evaluate blood glucose control overnight under closed- loop insulin delivery with MD-Logic Artificial Pancreas (MDLAP) system in patients with type 1 diabetes in the hospital settings,at diabetes camp settings and finally at patient's home .

Study Objectives To determine the safety and efficacy of using the MDLAP system to automatically control blood glucose in type 1 diabetic patients.

Study Scope This is a three center, prospective pilot trail to evaluate blood glucose control under closed-loop insulin delivery with MD-Logic Artificial Pancreas (MDLAP) system in patients with type 1 diabetes, being conducted in: Tel Aviv, Israel;Ljubljana, Slovenia and Hannover, Germany

Study will be consist from six segments:

In segment 1, 15 eligible patients will be enrolled for the pilot study. 5 patients will be recruited at each center.Data generated from the first patient at each center will not be included at the final statistical analysis and will be used to assess logistical and training issues only.

On the second segment, 54 eligible subjects will be enrolled (18 at each center). Each subject will participate in the two consecutive overnight sessions in diabetes camp settings, one under closed-loop with MDLAP and one under sensor augmented pump therapy. Staying at a camp, can represent the home setting, but has on site the support of a medical team trained in diabetes. A remote safety and control diabetes management system will be utilized at this segment to enable the supervising personnel to alert the patient and intervene in cases of impending hypoglycemia, long standing hyperglycemia and technical faults of any component of the AP system.

In the third segment,9-20 eligible patients will be enrolled at the Israeli center only.Each subject will participate in up to four consecutive overnight under closed loop with MDLAP and up to four additional overnight under regular sensor augmented pump therapy at home.In similar to segment 2, we will use also at segment 3 the remote safety and control diabetes management system which enable the supervising personnel to alert the patient or parents and intervene in cases of impending hypoglycemia, long standing hyperglycemia and technical faults of any component of the AP system.

On the fourth segment, 45-60 patients will be enrolled at the Israeli center only, This segment will be conducted at a diabetes camp and will consist of two main parts. In part 1, 15-20 patients will be randomized to participate in one of the two groups: 2-4 nights under closed loop control while the MD-Logic learning algorithm is activated or 2-4 nights under closed loop control without activating the MD-Logic learning algorithm. In part 2 of the forth segment 30-40 patients will participate in two consecutive 24-48 hours sessions,one under closed loop control and the second under sensor augmented pump therapy.

On the fifth segment 40-80 eligible patients will be enrolled at the Israeli center only and will be conducted at patient's home. This segment will consist of two main parts .The first 10 patients will participate in a pilot session and data gathered at this pilot session will not be used at the final analysis. At part 1 each subject will participate in 4 weeks-1.5 months period of over nights either using closed-loop with MDLAP or using sensor augmented pump (SAP) therapy.At the end of the first 4 weeks-1.5 months of the study, statistical analysis will be performed in order to decide whether to extend the study with an optional period of extra 4 weeks-1.5 months.In case it will be decided to extend the study, additional 4 weeks-1.5 months intervention period following completion of final visit activities will be offered to participants. Subjects that have participated in the control group (sensor augmented pump therapy) will be offered the opportunity to continue to 4 weeks-1.5 months of closed-loop control and the study group will be offered to switch to sensor augmented pump therapy. In segment 5 part 2, up to 40 patients will be enrolled. Each patient will participate in 3 months study period either using overnight closed loop under MDLAP or sensor augmented pump therapy. Participants in segment 5 part 2 will be offered to participate in part 2A. At this part, sleep quality assessment will be made (by using actigraf and sleep questionnaire). At the end of this period an optional 3 months extension period will be offered with the other arm (cross-over).

Segment 6 will be consist of two main parts.In part 1 up to 40 eligible patients will be enrolled at the Israeli center only. Each subject will participate in up to 72 hours of closed-loop with MDLAP at home and up to 72 hours under regular sensor augmented pump therapy . The sequence of the treatment intervention will be randomly assigned. In part 2 of this segment 40 eligible patients will enrolled at the Israeli center only. Each subject will participate in up to 2 weeks of closed loop with MDLAP at home and up to 2 weeks under regular sensor augmented pump therapy. The sequence of the treatment intervention will be randomly assigned

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes (>1yr since diagnosis)
* Insulin infusion pump therapy for at least 3 months
* Patients whom uses continuous glucose sensor for at least 2 weeks(for segment 5) or will undergo run-in period of 2 weeks of glucose sensor wear before continue to baseline assessment (only for patients participating at segment 3 and 4)
* Age ≥ 10 years until 65 years
* HbA1c at inclusion ≥ 6.5 and <10
* Patients willing to follow trail instructions
* Patients live with at least one other adult person (segment 3, 5, and 6 only)
* BMI Standard Deviation Score - below the 97th percentile for age(in segment 5 and 6 BMI SDS - below the 95th percentile for age)
* An internet connection at patient's home (only for patients participating at segment 3 and 6)
* Patients with care givers who are capable of operating a computer based system

Exclusion Criteria:

* Concomitant diseases that influence metabolic control
* Participation in any other interventional study
* Known or suspected allergy to trial products
* Any significant diseases or conditions including psychiatric disorders and substance abuse that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study, or compromise patient safety
* Diabetic ketoacidosis in the past 1 month.
* Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment.
* Current use of oral glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* Subject is participating in another drug or device study that could affect glucose measurements or glucose management.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of hypoglycemic events | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Number of overnight hypoglycemic events below 63 mg/dl, between bed time to 07:00
Time spent in hypoglycemia | final visit (day 26 for participants at segment 1 , day 14 for participants in segment 2 and day 20 for participants in segment 3, 4 weeks-1.5 months for participants in segment 5)
  Reduction of time spent in hypoglycemia defined as sensor glucose level below 60 mg/dL at segments 1&2 below 63 mg/dl at segment 3 and below 70 mg/dl in segment 5
Reduction in overnight mean glucose level | final visit (day 26 for participants at segment 1 and day 14 for participants in segment 2)
  Reduction in overnight mean glucose level
Increase in time spent in the target range | day 14 for participants in segment 4
  Increase in time spent in the target range defined as sensor glucose level within 63 to 140 mg/dl (3.5 to 7.8 mmol/l)
Increase in time spent in the target range of sensor glucose level within 70-180 mg/dl | day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
  Increase in time spent in the target range of sensor glucose level within 70-180 mg/dl
Sleep efficacy | final visit (after7 months for participants at segment 5 part 2A)
  Sleep efficacy as measured by Actigraph

SECONDARY OUTCOMES:
Percentage of time spent in the target range | final visit (day 26 for participants at segment 1 , day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Percentage of time spent in the target range,defined as sensor glucose level within 63 to 140 mg/dl (3.5 to 7.8 mmol/l)and between 70 to 140 mg/dl(3.9 to 7.8 mmol/L)
Percentage of time spent in the tight target range | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Percentage of time spent in the target range, defined as sensor glucose level within 80 to 120 mg/dl (3.5 to 7.8 mmol/l)
Average (SD) of blood glucose levels | final visit (day 26 for participants at segment 1and 4 and day 14 for participants in segment 2, day 20 for participants in segment 3, day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6)
  Average (SD) of blood glucose levels
Percentage of time spent below 60 mg/dl and below 70 mg/dl | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Percentage of time spent below 60 mg/dl and below 70 mg/dl
Percentage of time spent above 140, 180, 250 mg/dl (7.8, 10, 13.9 mmol/l) | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3 )
  Percentage of time spent above 140, 180, 250 mg/dl (7.8, 10, 13.9 mmol/l)
Glucose variability | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3 )
  Glucose variability
Control Variability Grid Analysis (CVGA) | final visit (day 26 for participants at segment 1 and day 14 for participants in segment 2)
  Control Variability Grid Analysis (CVGA)
number of accurate alerts related to the remote safety and control diabetes management system | final visit (day 26 for participants at segment 1 and day 14 for participants in segment 2)
  number of accurate alerts related to the remote safety and control diabetes management system
Number of hypoglycemic events below 60 and 70 mg/dl (3.3, 3.9 mmol/l) | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Number of hypoglycemic events below 60 and 70 mg/dl (3.3, 3.9 mmol/l)
Area under the curve <60,<63,<70,>140,>180,>250 mg/dl(3.3,3.5,3.9,7.8,10,13.9) | final visit (day 26 for participants at segment 1, day 14 for participants in segment 2 and 4 and day 20 for participants in segment 3)
  Area under the curve <60,<63,<70,>140,>180,>250 mg/dl(3.3,3.5,3.9,7.8,10,13.9)
• The percentage of nights mean overnight sensor glucose levels was within 90-140mg/dl (5-7.8 mmol/l) | final visit (day 14 ) for participants in segment 4 only
Postprandial peak blood glucose and 2 hours postprandial blood glucose (segment 4 and 6 only) | Final visit (day 14 ) for participants in segment 4 part 1, day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
Artificial Pancreas technical performance, defined as the total frequency of failures | Final visit (day 14 ) for participants in segment 4 only
  Artificial Pancreas technical performance, defined as The total frequency of failures (number of failures/night) of each following system components: sensor communication, pump communication, controller, user interface
Analysis of the number of sensor data point not received to the artificial pancreas device divided by the total number of possible data points to be received. | Final visit (day 14 ) for participants in segment 4 only
Percent time of active closed-loop control | Final visit (day 14) for participants in segment 4 only
  Percent time of active closed-loop control defined as the number of minutes the MD-Logic system was functioning properly (computation of insulin infusion, and insulin actually delivered) divided by the maximum number of minutes the MD-Logic system should have been active (as per protocol)
sensor accuracy | final visit (day 14 for participants in segment 4 only)
  comparison of paired data points between capillary glucose level and Continuous Glucose Monitoring
The time spent in hypoglycemia | After 4 weeks-1.5 month at segment 5 only (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  The time spent in hypoglycemia below 50 mg/dl (2.8 mmol/l).
The number of hypoglycemic events below 60 and 50 mg/dl | After 4 weeks- 1.5 months only at segment 5(in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  The number of hypoglycemic events below 60 and 50 mg/dl (event defined duration of at least 20 minutes).
The time sensor glucose level spent within 70 to 140 mg/dl (3.9 to 7.8 mmol/l) | After 4 weeks- 1.5 months only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
The time spent in hyperglycemia | After 4 weeks-1.5 monts only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  The time spent in hyperglycemia above 240 mg/dl (13.3 mmol/l).
Patient's diabetes treatment satisfaction | After 4 weeks-1.5 months only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  Patient's diabetes treatment satisfaction using Diabetes Treatment Satisfaction Questionnaire
Acceptance and use intention of an Artificial Pancreas | after 4 weeks- 1.5 months only at segment 5(in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  Acceptance and use intention of an Artificial Pancreas for participant and for parents
Fear of hypoglycemia | After 4 weeks- 1.5 months only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  Fear of hypoglycemia using questionaire
Satisfaction with Artificial Pancreas | After 4 weeks- 1.5 months only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
  Satisfaction with Artificial Pancreas using questionaire
Average percentage of overnight operation of the closed-loop control | After 4 weeks-1.5 months only at segment 5 (in addition after additional 4 weeks-1.5 months if segment 5 will be extended)
Percentage of time spent below 50, 60, 70 mg/dl | day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
  Percentage of time spent below 50, 60, 70 mg/dl
Number of hypoglycemic events below 50, 60, 70 mg/dl | day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
  Number of hypoglycemic events below 50, 60, 70 mg/dl
Percentage of time spent above 180, 250 mg/dl | day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
  Percentage of time spent above 180, 250 mg/dl
Number of readings below 70 mg/dl | day 20 for participants in segment 4 part 2 and day 56 for participants in segment 6
Automatic Caller System (ACS) technical performance and number of accurate alerts | final visit (after 7 months for participants at segment 5 part 2)
number of research team intervention | final visit (after 7 months for participants at segment 5 part 2)
HbA1c | final visit (after 7 months for participants at segment 5 part 2)
Number of awake bouts per night | final visit (after 7 months for participants at segment 5 part 2A)
  Number of awake bouts per night as measured by Actigraph
Total wake up time per night | final visit (after 7 months for participants at segment 5 part 2A
  Total wake up time per night as measured by Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schenider Children's Medical
Locations (3):
- Diabetes -Zentrum fuer kinder und jugendliche, Hanover, Germany
- Schneider Children's Medical center, Petah Tikva, Israel
- University Children's Hospital, Ljubljana, Slovenia

REFERENCES:
- [Derived] Biester T, Nir J, Remus K, Farfel A, Muller I, Biester S, Atlas E, Dovc K, Bratina N, Kordonouri O, Battelino T, Philip M, Danne T, Nimri R. DREAM5: An open-label, randomized, cross-over study to evaluate the safety and efficacy of day and night closed-loop control by comparing the MD-Logic automated insulin delivery system to sensor augmented pump therapy in patients with type 1 diabetes at home. Diabetes Obes Metab. 2019 Apr;21(4):822-828. doi: 10.1111/dom.13585. Epub 2018 Dec 21. PMID 30478937
- [Derived] Nimri R, Muller I, Atlas E, Miller S, Fogel A, Bratina N, Kordonouri O, Battelino T, Danne T, Phillip M. MD-Logic overnight control for 6 weeks of home use in patients with type 1 diabetes: randomized crossover trial. Diabetes Care. 2014 Nov;37(11):3025-32. doi: 10.2337/dc14-0835. Epub 2014 Jul 30. PMID 25078901
- [Derived] Nimri R, Danne T, Kordonouri O, Atlas E, Bratina N, Biester T, Avbelj M, Miller S, Muller I, Phillip M, Battelino T. The "Glucositter" overnight automated closed loop system for type 1 diabetes: a randomized crossover trial. Pediatr Diabetes. 2013 May;14(3):159-67. doi: 10.1111/pedi.12025. Epub 2013 Feb 28. PMID 23448393
- [Derived] Phillip M, Battelino T, Atlas E, Kordonouri O, Bratina N, Miller S, Biester T, Stefanija MA, Muller I, Nimri R, Danne T. Nocturnal glucose control with an artificial pancreas at a diabetes camp. N Engl J Med. 2013 Feb 28;368(9):824-33. doi: 10.1056/NEJMoa1206881. PMID 23445093